CLINICAL TRIAL: NCT06992128
Title: Romiplostim N01 Combined With Glucocorticoids as the First-line Treatment for Newly Diagnosed Adult Primary Immune Thrombocytopenia (ITP): A Multicenter, Interventional Trial
Brief Title: Romiplostim N01 Combined With Glucocorticoids as the First-line Treatment for Newly Diagnosed Adult Primary Immune Thrombocytopenia: A Multicenter, Interventional Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Weifang People's Hospital (Other); Shenzhen Second People's Hospital (Other); The Affiliated Hospital of Qingdao University (Other); The Affiliated Hospital of Nantong University (Unknown); The First Affiliated Hospital of Bengbu Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Changzhi Medical College (Other); North China University of Science and Technology (Other); Tianjin Hospital of ITCWM-Nankai Hospital (Unknown); Baoding First Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-ITP-IIT-001
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: ITP; Romiplostim; Continuous Remission; First-line Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- romiplostim N01 combined with glucocorticoids (Experimental)
  Interventions: Drug: Romiplostim N01 combined with dexamethasone
- glucocorticoids (Active Comparator)
  Interventions: Drug: Dexamethasone monotherapy

INTERVENTIONS:
Drug: Romiplostim N01 combined with dexamethasone — Dexamethasone (HD-DXM) at a dose of 40mg/d for 4 days constitutes one cycle. If there is no response on the 10th day, repeat it once. The administration can be either oral or intravenous. Meanwhile, romiplostim N01 is administered with an initial dose of 3µg/kg by subcutaneous injection within 4 days of dexamethasone treatment once a week for up to 6 months.
  Arms: romiplostim N01 combined with glucocorticoids
Drug: Dexamethasone monotherapy — Dexamethasone (HD-DXM) 40mg/d × 4 days, one cycle. If there is no response on the 10th day, repeat once, administered either orally or intravenously.
  Arms: glucocorticoids

SUMMARY:
This prospective, multicenter, randomized study aim to evaluate the efficacy and safety of romiplostim N01 combined with glucocorticoids as the first-line treatment for newly diagnosed adult primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The primary endpoint of this study is to assess the efficacy of romiplostim N01 combined with glucocorticoids in untreated newly diagnosed adult ITP patients after 6 months of administration. 129 eligible subjects were randomized to either romiplostim N01 combining glucocorticoids or glucocorticoids treatment in 2:1 ratio. Administration protocol: Experimental group: Dexamethasone (HD-DXM) 40mg/d × 4d, one cycle. If there is no response on the 10th day, repeat once, administered orally or intravenously. Simultaneously, romiplostim N01 is administered, with an initial dose of 3µg/kg, by subcutaneous injection once a week, for up to 6 months. Control group: Dexamethasone (HD-DXM) 40mg/d × 4d, one cycle. If there is no response on the 10th day, repeat once, administered orally or intravenously. The initial dose of romiplostim N01 administration was 3µg/kg and can be initiated within 4 days of dexamethasone treatment. The dose of romiplostim N01 was adjusted according to the subject platelet count during the treatment period. When the platelet count is < 50 × 10^9/L, the patient will receive an increment in the dose of romiplostim N01 by 2µg/kg weekly, with a maximum dose of 10µg/kg. When 200 × 10^9/L > platelet count ≥ 50 × 10^9/L, the administration dosage remains unchanged. When 400 × 10^9/L > platelet count ≥ 200 × 10^9/L for two consecutive weeks, the dose is reduced by 1µg/kg. When the platelet count is ≥ 400 × 10^9/L, discontinue the drug. When the platelet count < 200 × 10^9/L, resume administration, and the administration dose is 1µg/kg less than before drug cessation. All subjects were followed up until the 24th week after the end of treatment through clinical follow-up or telephone follow-up. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events, concomitant medications and concomitant treatments are also recorded throughout the study. The researcher can increase the number of visits as necessary for AE follow-up to monitor the alleviation of AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the written informed consent form before enrollment;
2. Age ranging from 18 to 75 years old;
3. Be clinically diagnosed with primary immune thrombocytopenia for less than 3 months before randomization;
4. have not received any prior treatments for ITP.
5. Have not received romiplostim treatment;
6. ECOG PS score: 0 - 2;
7. Platelet value < 30×10^9/L;
8. The expected survival period at the screening is ≥ 12 weeks;
9. For subjects of reproductive age, agree to take reliable contraceptive measures throughout the study period (including male or female condoms, contraceptive foams, contraceptive gels, contraceptive membranes, contraceptive ointments, contraceptive suppositories, abstinence, and intrauterine device placement, etc.); Female subjects who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation or menopause for more than 1 year, and male subjects who have undergone bilateral vasectomy or ligation are excluded;
10. Voluntarily join this study, sign the informed consent form, and have good compliance.

Exclusion Criteria:

1. Suffering from other secondary thrombocytopenia except ITP, including but not limited to leukemia, thrombocytopenia caused by tumor treatment, myeloproliferative diseases, multiple myeloma, myelodysplastic syndrome, common variable immunodeficiency, and hereditary thrombocytopenia, etc.;
2. Having undergone splenectomy before the first administration;
3. Having received ITP drug treatment (including emergency treatment) before the first administration;
4. Having used drugs with c-Mpl (thrombopoietin receptor) stimulating effects within 4 weeks before the first administration;
5. Having received hematopoietic growth factor preparations (such as granulocyte colony-stimulating factor, macrophage colony-stimulating factor, erythropoietin, interleukin-11, etc.) within 4 weeks before the first administration;
6. Having received antibody drugs (such as rituximab, etc.) within 14 weeks before the first administration;
7. Having received any Chinese herbal medicine or nutritional supplement (except vitamin supplements and mineral supplements) for the purpose of increasing platelets within 1 week before the first administration;
8. Having been diagnosed with arterial thrombosis (such as cerebral thrombosis, transient ischemic attack or myocardial infarction), or having a history or complication of venous thrombosis (such as deep vein thrombosis, pulmonary embolism), or using anticoagulants or antiplatelet drugs at the beginning of screening;
9. Having a history of severe cardiovascular diseases (such as grade III/IV congestive heart failure, arrhythmia or angina pectoris that increases the risk of thromboembolic events, unstable angina pectoris, having undergone coronary artery stent implantation, angioplasty or coronary artery bypass grafting);
10. Secondary thrombocytopenia caused by autoimmune diseases such as antiphospholipid antibody syndrome, systemic lupus erythematosus, Hashimoto's thyroiditis, Even's syndrome and Sjogren's syndrome;
11. Positive results for either human immunodeficiency virus antibody or syphilis antibody screening; positive hepatitis C antibody and HCV-RNA exceeding the upper limit of the study center's laboratory test; positive hepatitis B surface antigen and HBV-DNA exceeding the upper limit of the study center's laboratory test;
12. Having participated in other clinical studies within 3 months before the first administration;
13. Being pregnant or lactating, or having a pregnancy plan;
14. Having fertility and being judged by the researcher as not fully adopting contraceptive measures;
15. Having a history of severe drug allergic reactions or being known to be allergic to glucocorticoids or Nplate® (romiplostim) or the components of QL0911;
16. Unable to comply for mental reasons;
17. Judged by the researcher as not suitable to participate in this trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-05-22 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with continuous remission | 6 months
  Continuous remission is defined as the maintenance of the therapeutic effect of patients for at least 6 months since achieving remission, without the need for additional ITP-specific treatment.

SECONDARY OUTCOMES:
The total effective rate OR | 6 months
  The total effective rate OR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Response R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms).
The proportion of patients with the initial response (reaching the effective standard within one month of the start of treatment) | one month of the start of treatment
  The total effective rate OR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Response R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within one month).
The proportion of patients reaching the effective standard 3 months after the start of treatment | 3 months after the start of treatment]
  The total effective rate OR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Response R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within 3 month).
The proportion of patients reaching the effective standard 6 months after the start | 6 months after the start of treatment
  The total effective rate OR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Response R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within 6 month).
The proportion of patients reaching the effective standard 9 and 12 months after the start of treatment | 9 and 12 months after the start of treatment
  The total effective rate OR = CR + R (Complete response CR, platelet count ≥ 100×10^9/L, and no bleeding symptoms; Response R, platelet count is between 30×10^9/L and 100×10^9/L, and at least doubles compared to the baseline value, and no bleeding symptoms within 9 and 12 month).
The maximum consecutive weeks of platelet response | 6 months
  The consecutive weeks with platelet count > 30×10^9/L in the absence of any rescue treatment.
The proportion of subjects receiving rescue treatment. | 6 months
  The proportion of subjects receiving rescue treatment.
According to the WHO bleeding score standard, the incidence and severity of bleeding symptoms. | 6 months
  According to the WHO bleeding score standard, the incidence and severity of bleeding symptoms
The incidence of adverse events | 6 months
  Evaluated using Version 5.0 of the "Common Terminology Criteria for Adverse Events (NCI CTC AE)".

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No